CLINICAL TRIAL: NCT00934466
Title: A Randomized Clinical Trial to Assess the Effects of Single Doses of MK2637 and Dextromethorphan on Cerebral Cortex Excitability in Healthy Subjects
Brief Title: Study of the Effect of Single Doses of MK2637 and Dextromethorphan on Cerebral Cortex Excitability (2637-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2637-008; MK2637-008; 2009_608
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): MK2637 120 mg
  Interventions: Drug: MK2637
- 2 (Experimental): MK2637 50 mg
  Interventions: Drug: Comparator: MK2637
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 4 (Active Comparator): Dextromethorphan 220 mg
  Interventions: Drug: Comparator: Dextromethorphan
- 5 (Active Comparator): Dextromethorphan 110 mg
  Interventions: Drug: Comparator: Dextromethorphan

INTERVENTIONS:
Drug: MK2637 — Single dose of 120 mg MK2637 capsules in one of five treatment periods.
  Arms: 1
Drug: Comparator: MK2637 — Single dose of 50 mg MK2637 capsules in one of five treatment periods.
  Arms: 2
Drug: Comparator: Placebo — Single dose of placebo only in one of five treatment periods.
  Arms: 3
Drug: Comparator: Dextromethorphan — Single dose of 220 mg dextromethorphan capsules in one of five treatment periods.
  Arms: 4
Drug: Comparator: Dextromethorphan — Single dose of 110 mg dextromethorphan capsules in one of five treatment periods.
  Arms: 5

SUMMARY:
This study will assess transcranial magnetic stimulation (TMS) as a biomarker and characterize TMS readouts of the activity of MK2637 and dextromethorphan. Resting quantitative electroencephalography(qEEG) readouts are also characterized with MK2637 and dextromethorphan.

ELIGIBILITY:
Inclusion Criteria:

* Subject is right-handed
* Subject is in good health
* Subject is a nonsmoker

Exclusion Criteria:

* Subject works a night shift
* Subject has a history of any illness that might make participation in the study unsafe or confound the study results
* Subject has a history of head injury

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Increase in Motor Evoked Potential (MEP) after dosing with dextromethorphan compared to placebo | 5 Hours after initial dosing
Increase in amplitude in the gamma frequency band (24-60 Hz) of resting qEEG after dosing with dextromethorphan compared to placebo | 4 Hours after initial dosing

SECONDARY OUTCOMES:
Increase in amplitude in the theta frequency band (4-8 Hz) of resting qEEG after dosing with MK2637 compared to placebo | 6.5 hours after initial dosing
Change in Motor Evoked Potential (MEP) after dosing with MK2637 as compared to placebo | 5 hours after initial dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC